CLINICAL TRIAL: NCT05750394
Title: Cesarean 123 Trial: Prospective Randomized Trial Comparing Single, Double and Triple Layer Uterine Closures During Cesarean Delivery
Brief Title: Cesarean 123 Trial: Randomized Trial Comparing Single, Double and Triple Layer Uterine Closures During Cesarean Delivery
Acronym: C123T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, James Greenberg, MD, Vice Chair OB/GYN, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P000041
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy Related
Keywords: Cesarean; Myometrium; scar thickness; niche
MeSH Terms: interventions — Endomet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Radiologist blinded to closure method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Single Layer Closure (Active Comparator): Single layer closure using the following technique:
  a. Closure of the myometrium and serosa with one (1) 0 V-Loc 90 suture on a GS-24 needle using an unlocked technique. The endometrium should be excluded.
  Interventions: Procedure: Uterine layers closed; Device: Suture Type; Procedure: Endometrium
- Double Layer Closure (Active Comparator): Double layer closure using the following technique:
  1. Closure of the full thickness of the myometrium with one (1) Monocryl suture on a CT needle using a running locked technique. The endometrium should be excluded.
  2. Imbrication of the first layer with one (1) Monocryl suture on a CT needle using a running un-locked technique
  Interventions: Procedure: Uterine layers closed; Device: Suture Type; Procedure: Endometrium
- Triple Layer Closure (Active Comparator): Triple layer closure of Endometrium, Myometrium and Serosa (EMS) using one of the the following two techniques:
  1. Closure of the endometrium and 2-4 mm of internal myometrium with one (1) 2-0 V-Loc 90 suture on a GS-21 needle using an unlocked technique
  2. Closure of the remaining myometrium and serosa with one (1) 0 V-Loc 90 suture on a GS-24 needle using an unlocked technique
  or
  1. Closure of the endometrium and 2-4 mm of internal myometrium with one (1) 2-0 V-Loc 90 suture on a GS-21 needle using an unlocked technique
  2. Closure of the remaining myometrium with one (1) 0 V-Loc 90 suture on a GS-24 needle using an unlocked technique
  3. Closure of the serosa with one (1) 2-0 V-Loc 90 suture on a GS-21 needle using an unlocked technique
  Interventions: Procedure: Uterine layers closed; Device: Suture Type; Procedure: Endometrium

INTERVENTIONS:
Procedure: Uterine layers closed — Uterus closed with 1, 2 or 3 layers
Device: Suture Type — Barbed or smooth
Procedure: Endometrium — Included or excluded

SUMMARY:
The goal of this clinical trial is to compare post-operative uterine scar thickness in people who have had the uterus closed during cesarean sections by one of three different methods. The main questions it aims to answer are:

* Residual myometrial thickness at the scar site assessed by MRI performed 4 months after the procedure
* Myometrial niche formation assessed by MRI performed 4 months after the procedure
* Scar healing ratio (HR) difference as defined by HR= residual myometrial thickness/total myometrial thickness
* Post-operative change in hemoglobin
* Time required for hysterotomy closure
* The number of extra sutures required to achieve surgeon-acceptable hemostasis

Participants undergoing scheduled cesarean sections will be randomized to one of three different uterine closure methods. The methods are:

1. Single layer closure using the following technique: Closure of the myometrium and serosa with one barbed suture using a running unlocked technique. The endometrium should be excluded.
2. Double layer closure using the following technique: Closure of the full thickness of the myometrium with one smooth suture using a running locked technique. The endometrium should be excluded. Followed by imbrication of the second layer with one smooth suture using a running unlocked technique.
3. Triple layer closure of Endometrium, Myometrium and Serosa (EMS) using one of the the following two techniques: Closure of the endometrium and 2-4 mm of internal myometrium with one barbed suture using a running unlocked technique followed by closure of the remaining myometrium and serosa with one barbed suture using a running unlocked technique. Or, Closure of the endometrium and 2-4 mm of internal myometrium with one barbed suture on using a running unlocked technique followed by closure of the remaining myometrium with one barbed suture a running unlocked technique followed by closure of the serosa with one barbed suture using a running unlocked technique.

Four months after the surgery, participants will have a MRI of the pelvis to assess the scar on the uterus.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Singleton gestation
* Nonurgent primary or secondary cesarean delivery at greater than 35w6d
* Body Mass Index (BMI) <35 kg/m^2

Exclusion Criteria:

* More than 1 prior cesarean delivery
* Multiple gestation
* Known coagulation disorder or current use of anti-coagulants
* Mullerian anomalies
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant people having cesarean delivery
Enrollment: 120 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Myometrial thickness | 4 months
  Residual myometrial thickness at the scar site assessed by MRI performed

SECONDARY OUTCOMES:
Niche | 4 months
  Myometrial niche formation assessed by MRI performed
Scar ratio | 4 month
  Scar healing ratio (HR) difference as defined by HR= residual myometrial thickness/total myometrial thickness by MRI
Blood loss | 1 day
  Post-operative change in hemoglobin
Time for closure | Immediate
  Time required for hysterotomy closure
Extra sutures | Immediate
  The number of extra sutures required to achieve surgeon-acceptable hemostasis

CONTACTS AND LOCATIONS:
Overall Officials: James A. Greenberg, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion

REFERENCES:
- [Result] Roberge S, Demers S, Girard M, Vikhareva O, Markey S, Chaillet N, Moore L, Paris G, Bujold E. Impact of uterine closure on residual myometrial thickness after cesarean: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):507.e1-507.e6. doi: 10.1016/j.ajog.2015.10.916. Epub 2015 Nov 11. PMID 26522861
- [Result] Alessandri F, Evangelisti G, Centurioni MG, Gustavino C, Ferrero S, Barra F. Fishbone double-layer barbed suture in cesarean section: a help in preventing long-term obstetric sequelae? Arch Gynecol Obstet. 2021 Sep;304(3):573-576. doi: 10.1007/s00404-021-06121-8. PMID 34146146